CLINICAL TRIAL: NCT00752492
Title: Acceleration of Recovery From General Anesthesia - Efficacy of Isocapnic Hyperpnoea in Obese Patients Undergoing Isoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Rita Katznelson, Toronto General Hospital, University Health Network
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UHNREB08-0019B
Record Dates: First submitted 2008-07-22; First posted 2008-09-15 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Recovery Time From Isoflurane Anesthesia in Obese Patients
Keywords: Isocapnic hyperpnoea; obesity; isoflurane; Recovery of obese patient from isoflurane anesthesia
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study intervention (Active Comparator): Patient will be disconnected from the anesthetic circuit and connected to the resuscitation bag attached to the IH system. Ventilation will be assisted to maintain tidal volume of 8-10 mL/kg and respiratory rate of 20-25 breaths per minute to achieve minute ventilation of 15-20 L/min. Isocapnia manifold will maintain end-tidal PCO2 in range of 40-50 mm Hg.
  Interventions: Other: Isocapnic Hyperpnoea

INTERVENTIONS:
Other: Isocapnic Hyperpnoea — IH is a method of increasing alveolar ventilation (Va) while preventing the unwanted hypocapnia by addition of CO2 to the inhaled mixture.

SUMMARY:
Faster recovery from anesthesia is important for obese patients because they are at high risk of respiratory complications following tracheal extubation. Isoflurane has several properties that make it a preferable agent for anesthesia in obese patients. Its main limitation is a longer recovery time due to slower elimination in comparison to other agents. Elimination of isoflurane from the lungs can be accelerated by increasing in patient's minute ventilation, which decreases the level of CO2 in blood (hypocapnia).Isocapnic Hyperpnoea (IH) is a method allowing increased ventilation and therefore enhancement of the elimination of inhalation agents while maintaining a normal blood CO2 level. The investigators will compare recovery time from isoflurane anesthesia in obese patients during standard anesthesia management protocol (control) to a group treated with IH.

ELIGIBILITY:
Inclusion Criteria:

Elective gynecological or urological procedure,

* BMI > 35 kg/m²,
* ASA I-III,
* Signed informed consent.

Exclusion Criteria:

* Lack of informed consent,
* ASA IV-V,
* Contra-indications to isoflurane anesthesia or other anesthetics included in the protocol,
* History of cardiac or respiratory disease,
* Alcohol or drug abuse,
* Psychiatric illness and/or medications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Time from the end of anesthesia (turning isoflurane vaporizer off) to the readiness for Post Anesthesia Care Unit (PACU) discharge. | Intraoperatively and Post Anesthetic Care Unit

SECONDARY OUTCOMES:
Times from end of anesthesia to BIS exceeds 75, b) eye-opening to verbal command, c) extubation, d) readiness for leaving | Intraoperatively and Post Anesthetic Care Unit
Sedation/Pain scores in the PACU. | Intraoperatively and Post Anesthetic Care Unit
Change in exhaled isoflurane concentrations in the 1st hour postoperatively. | Intraoperatively and Post Anesthetic Care Unit

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada